CLINICAL TRIAL: NCT04997356
Title: Computer-Based Cognitive Games, Personality, and Behavior Study
Brief Title: Hostile Bias Modification Training (HBMT) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2637
Record Dates: First submitted 2021-07-29; First posted 2021-08-09 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Anger; Stress; Aggression
MeSH Terms: conditions — Aggression

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are blinded to study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hostile Bias Modification (HBM) Training plus Unambiguous Feedback (Experimental): Volunteers will complete a novel computer-based hostile bias modification training where they are instructed to respond to word fragments (words with missing letters) based on whether the word fragments can be completed to form aggressive or positive/neutral words. They are instructed not to respond if only an aggressive word can be formed. They will receive unambiguously hostile feedback to an essay.
  Interventions: Behavioral: Hostile Bias Modification Training
- Other training plus Unambiguous Feedback (Placebo Comparator): Volunteers will complete a computer-based task where they are instructed to respond to word fragments (words with missing letters) regardless of whether the fragments can make hostile or ambiguous words. They will receive unambiguously hostile feedback to an essay.
  Interventions: Behavioral: Other training
- Hostile Bias Modification (HBM) Training plus Ambiguous Feedback (Experimental): Volunteers will complete a novel computer-based hostile bias modification training where they are instructed to respond to word fragments (words with missing letters) based on whether the word fragments can be completed to form aggressive or positive/neutral words. They are instructed not to respond if only an aggressive word can be formed. They will receive ambiguously hostile feedback to an essay.
  Interventions: Behavioral: Hostile Bias Modification Training
- Other training plus Ambiguous Feedback (Placebo Comparator): Volunteers will complete a computer-based task where they are instructed to respond to word fragments (words with missing letters) regardless of whether the fragments can make hostile or ambiguous words. They will receive ambiguously hostile feedback to an essay.
  Interventions: Behavioral: Other training

INTERVENTIONS:
Behavioral: Hostile Bias Modification Training — Volunteers will complete a novel computer-based hostile bias modification training where they are instructed to respond to word fragments (words with missing letters) based on whether the word fragments can be completed to form aggressive or positive/neutral words. They will refrain from making words that can only form aggressive words.
  Other Names: HBMT
  Arms: Hostile Bias Modification (HBM) Training plus Ambiguous Feedback; Hostile Bias Modification (HBM) Training plus Unambiguous Feedback
Behavioral: Other training — Volunteers will complete a computer-based task where they are instructed to respond to word fragments (words with missing letters) regardless of whether the fragments can make hostile or ambiguous words.
  Arms: Other training plus Ambiguous Feedback; Other training plus Unambiguous Feedback

SUMMARY:
The primary objective of the present protocol is to evaluate the effectiveness of real HBMT versus placebo on reducing HAB and aggression.

The secondary objectives of the present protocol are:

1. Investigate the role of individual difference variables on HAB, interpersonal aggression, and effects of HBMT.
2. Collect vocal recording data to inform the development of algorithms to predict emotional stress from changes in speech.

DETAILED DESCRIPTION:
Aggression refers to causing harm to someone who is motivated to avoid that harm (Anderson & Bushman, 2002). Many Soldiers report heightened levels of anger and display elevated rates of aggressive behavior following combat deployments (Adler et al., 2011; Jakupcak et al., 2007; Novaco & Chemtob, 2015; Orth & Wieland, 2006; Thomas et al., 2010). Treating and addressing anger and aggression in combat Veterans can improve Soldier health as well as promote force readiness and lethality. One key predictor of anger and aggression when responding to the actions of other people is the extent to which the victim believes that the provocateur acted in an intentionally hostile manner (e.g., being shoved on purpose) versus not intending to be hostile (e.g., being shoved by mistake; De Castro, Veerman, Koops, Bosch, & Monshouwer, 2002). This is called "hostile attributional bias" (HAB). Interpretation and attribution biases toward perceiving threats and danger are elevated in individuals with posttraumatic stress symptoms (Bonyea, Johnson, and Lang, 2017).

In the present study, the investigators test the effectiveness of a computer-based training called Hostile Bias Modification Training (HBMT) to reduce HAB and aggressive behavior in response to an ambiguous provocation (ambiguously hostile comments). Volunteers will complete a real or placebo version of a computer training designed to reduce HAB, then receive and react to either unambiguously hostile or ambiguously hostile feedback. The feedback is in regards to an essay the volunteer was asked to write as part of the study. The investigators predict that receiving the real (vs. placebo) computer training will reduce HAB in response to the ambiguous feedback, but not the unambiguous feedback. Volunteers will then partake in a second computer task, which involves a reaction time competition against the same confederate where the loser receives a penalty in the form of a short, unpleasant, acoustic tone delivered via headphones. The volunteer is told they can set the volume and duration of unpleasant acoustic tones that would be administered to the confederate. Aggression is operationalized as setting higher volumes and/or longer durations for tones. This will allow us to measure how aggressive volunteers are in response to ambiguous provocations and determine if the computer training is effective in reducing aggression to ambiguous provocations and if reduced HAB is the underlying mechanism of this effect. Finally, volunteers will complete a set of personality measures so we can determine if the effects of the computer training are contingent on individual differences. If successful, this research would add validity to a potential intervention to help people suffering from anger and aggression management issues to reduce their symptoms.

The investigators are also using this experiment as an opportunity to collect vocal pattern data to inform the development of algorithms to predict emotional stress from changes in vocal patterns. As such, voice recordings of volunteers reading standardized scripts will be made at three points in the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female, ages 18-39 (inclusive)
* Must confirm when asked by the experimenter that they are of normal hearing without the use of a hearing aid or have been diagnosed with any condition that produces a strong sensitivity to sound (e.g., misophonia, hyperacusis) to the best of their knowledge.
* Must be able to provide written informed consent before commencing with experimental procedures and perform experimental writing and reading tasks (i.e., must be able to fluently read/write in English).
* Must demonstrate satisfactory comprehension of the Informed Consent Document (ICD) by achieving a score of 100% correct on a short multiple-choice quiz .

Exclusion Criteria:

* not between ages 18-39
* not able to read/write fluently in English
* not of normal hearing without use of a hearing aid
* have been diagnosed with any condition that produces a strong sensitivity to sound (e.g., misophonia, hyperacusis)

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Essay Feedback Questionnaire | average of 30 minutes post-intervention
  8-item self-reported hostile attribution bias to ambiguously hostile or unambiguously hostile feedback (0-4). Higher scores indicate more bias.
Taylor Aggression Paradigm (TAP) | average of 45 minutes post-intervention
  The TAP objectively elicits and measures participant's aggression in response to provocation from an opponent. Aggression is operationalized as setting higher volumes and/or longer durations for tones (0-10). Higher scores indicate more aggression.

CONTACTS AND LOCATIONS:
Overall Officials: Margeaux V Auslander, PhD, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- Walter Reed Army Institute of Research, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-08-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT04997356/ICF_000.pdf